CLINICAL TRIAL: NCT04626622
Title: Kagocel for Oral Administration for the Prevention of Influenza and Other Acute Respiratory Viral Diseases in Young People
Brief Title: Kagocel® for the Prevention of ARVI and Influenza in Young People
Status: Completed | Type: Observational
Sponsor: Nearmedic Plus LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: version 1.0 from 21.11.2017
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Acute Upper Respiratory Tract Infection; Influenza; Respiratory Viral Infection
Keywords: Influenza; Acute Upper Respiratory Tract Infection; acute respiratory viral infection; ARVI; flu; cold; AURI
MeSH Terms: conditions — Influenza, Human; Common Cold

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ARVI and influenza prophylaxis with Kagocel (n=50): Prophylaxis according to routine practice and instructions for medical use of Kagocel.
  Group of patients receiving Kagocel for prevention of ARVI and influenza
  Interventions: Drug: Kagocel
- ARVI and influenza prophylaxis without any antiviral medicines (n=25): Group of patients receiving no any antiviral medicines for prevention of ARVI and influenza
  Interventions: Drug: No one

INTERVENTIONS:
Drug: Kagocel — Investigators could prescribe other drugs in frame of routine clinical practice
  Groups: ARVI and influenza prophylaxis with Kagocel (n=50)
Drug: No one — Investigators don't prescribe any antiviral drugs in frame of routine clinical practice
  Groups: ARVI and influenza prophylaxis without any antiviral medicines (n=25)

SUMMARY:
This study evaluates the use of Kagocel for the prevention of acute respiratory viral infections (ARVI) and influenza during the epidemic rise in the incidence of diseases in Russia in 2018 (epidemiology: the number of cases during the period of Kagocel administration and follow-up, bacterial exacerbations, the number of repeated episodes (reinfection), demographics of patients, safety, adherence to treatment) in students at risk due to stress, lack of sleep and fatigue.

DETAILED DESCRIPTION:
This non-interventional prospective study included 75 health students over the age of 18 who had no symptoms of acute respiratory viral infections (ARVI) and influenza at the time of inclusion and had not taken any antiviral medications to prevent ARVI and influenza for 30 days before.

The total duration of the study was 2 months: the first month participants took either Kagocel (the main group), or did not take anything at all (the control group), during the next 1 month all participants were monitored.

The diagnosis of influenza and ARVI has been confirmed in accordance with the world health organization (WHO) guidelines for the pharmacological treatment of pandemic influenza A (H1N1) 2009 and other influenza viruses. All patient examinations are conducted in accordance with local routine clinical practice and local and international standards of care.

By the study were analysed and compared those data between groups:

* demography
* anamnesis data (the incidence of ARVI and flu for previous year, the date of the lastest episode of the disease, the presence of concomitant diseases, including ENT-organs, the date of the lastest influenza vaccination).
* timelines: start of Kagocel's prevention - only for the group receiving Kagocel's prevention; start of the disease; duration of ARVI and influenza symptoms (fever, headache, runny nose, sore throat, cough); start of treatment
* symptomatic therapy (Yes/no, drug name)
* bacterial exacerbations (Yes/no)
* treatment of bacterial exacerbations (Yes/no)
* adverse events

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent to participate in the study.
* age from 18 to 30 years.
* the subject of the study does not have symptoms of ARVI and influenza at the time of inclusion in the study.
* there are no contraindications to the use of Kagocel: pregnancy and lactation, hypersensitivity to the components of the drug, lactase deficiency, lactose intolerance, glucose-galactose malabsorption (only for the group receiving kagocel prevention).
* the subject of the study should not to take other medications to prevent colds and flu while participating in the study.
* no history of participation in a clinical trial of any drug less than 30 days prior to inclusion in this study.
* no history of treatment by interferon or interferon inducers less than 30 days prior to inclusion in this study.

Exclusion Criteria:

* no exclusion criteria except participating in a current clinical trial because of non-interventional study design

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The young people over the age of 18 who had no symptoms of acute respiratory viral infections (ARVI) and influenza at the time of inclusion and had not taken any antiviral medications to prevent ARVI and influenza than 30 days prior to inclusion in this study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Total number of participants with ARVI or influenza | for the entire study period (for 2 months: for the 1st month of taking Kagocel+ for 1 month of follow-up after the end of the course of prevention)
Index of preventive efficacy | for the entire study period (for 2 months: for the 1st month of taking Kagocel+ for 1 month of follow-up after the end of the course of prevention)
  Index of preventive efficacy or I I= P2/P1; P1 - patients (who get disease; %) in the experimental (main) group; P2 - patients (who get disease; %) in the control group.
Total number of participants who required antibiotic therapy | for the entire study period (for 2 months: for the 1st month of taking Kagocel+ for 1 month of follow-up after the end of the course of prevention)

SECONDARY OUTCOMES:
Number of participants who have been ill repeatedly (twice or more) ARVI or influenza (reinfection) | for the entire study period (for 2 months: for the 1st month of taking Kagocel+ for 1 month of follow-up after the end of the course of prevention)
Number of vaccinated and not vaccinated participants who have ARVI or influenza | for the entire study period (for 2 months: for the 1st month of taking Kagocel+ for 1 month of follow-up after the end of the course of prevention)
Index of preventive efficacy for vaccinated participants | for the entire study period (for 2 months: for the 1st month of taking Kagocel+ for 1 month of follow-up after the end of the course of prevention)
  Index of preventive efficacy or I 1 I= P2/P1; P1 - patients (who get disease; %) in the experimental (main) group; P2 - patients (who get disease; %) in the control group.
Index of preventive efficacy for not vaccinated participants | for the entire study period (for 2 months: for the 1st month of taking Kagocel+ for 1 month of follow-up after the end of the course of prevention)
  Index of preventive efficacy or I 2 I= P2/P1; P1 - patients (who get disease; %) in the experimental (main) group; P2 - patients (who get disease; %) in the control group.
Number of vaccinated and not vaccinated participants who required antibiotic therapy | for the entire study period (for 2 months: for the 1st month of taking Kagocel+ for 1 month of follow-up after the end of the course of prevention)
Number of participants with treatment-related adverse events (AE) with regards to type and severity of AE (mild, moderate, severe; according to physician's opinion) | for the entire study period (for 2 months: for the 1st month of taking Kagocel+ for 1 month of follow-up after the end of the course of prevention)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Tikhonova, Dr. habilitated, Professor, Principal Investigator — Department of infectious diseases and epidemiology of Krasnoyarsk State Medical University named after Prof. V.F.Voino-Yasenetsky
Locations (1):
- Krasnoyarsk State Medical University, Krasnoyarsk, Krasnoyarsk Region, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Currently, great attention is paid to prevention of influenza and acute respiratory viral infections (ARVI). This article considers results of prospective observational study in prevention of influenza and ARVI among physicians [Publication on russian] — https://www.lvrach.ru/2018/10/15437102